CLINICAL TRIAL: NCT00751972
Title: Evaluation of the HeartWare Left Ventricular Assist Device for the Treatment of Advanced Heart Failure
Acronym: ADVANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HW003
Record Dates: First submitted 2008-09-10; First posted 2008-09-12 (Estimated); Results first posted 2014-05-02 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HeartWare® VAS (Experimental): Ventricular Assist Device (HeartWare® VAS)
  Interventions: Device: HeartWare® VAS

INTERVENTIONS:
Device: HeartWare® VAS — The HeartWare® LVAD is an implantable centrifugal pump that was designed to provide flows up to 10 L/min in a small device which is both lightweight and simple to use.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the HeartWare® LVAD System in patients listed for cardiac transplantation with refractory, advanced heart failure at risk of death. The primary endpoint is survival at 180 days which is defined as alive on the originally implanted HeartWare® LVAD or transplanted or explanted for recovery. Patient must survive 60 days post-explant for recovery to be considered successful. Secondary endpoints include:

* Overall survival
* Incidence of all serious adverse events, neurocognitive status and unanticipated adverse device effects.
* Incidence of all device failures and device malfunctions
* Quality of Life improvement, as measured by Kansas City Cardiomyopathy Questionnaire (KCCQ) and EuroQoL EQ-5D
* Functional status improvement, as measured by the New York Heart Association (NYHA) and 6-minute walk

The HeartWare® LVAD System was approved by the US FDA on November 20, 2012 as a bridge to cardiac transplantation (reference PMA P100047). Patients enrolled into this study will be followed to an outcome at six months, and then patients will receive continued follow-up in a separate study.

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 18 years of age at enrollment.
2. Body Surface Area (BSA) greater than or equal to 1.2 m2.
3. Patient is NYHA Class IV
4. Patient listed for cardiac transplantation
5. Patient meets United Network for Organ Sharing (UNOS) Status 1A or 1B listing criteria.
6. HeartWare® LVAD implant is planned as a bridge to transplant
7. The patient or legally authorized representative has signed the informed consent form

Exclusion Criteria:

1. Existence of any ongoing mechanical circulatory support (MCS) other than an intra-aortic balloon pump (IABP)
2. Prior cardiac transplant.
3. History of confirmed, untreated abdominal or thoracic aortic aneurysm > 5 cm.
4. Cardiothoracic surgery within 30 days of enrollment.
5. Acute myocardial infarction within 14 days of implant as diagnosed by ST or T wave changes on the ECG, diagnostic biomarkers, ongoing pain and hemodynamic abnormalities as described (Figure 2) in the guidelines published in ACC/AHA 2007 Guidelines for the Management of Patients with Unstable Angina/Non-ST-Elevation Myocardial Infarction; A Report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. JACC Vol. 50, No.7, 2007.
6. On ventilator support for > 72 hours within the fours days immediately prior to enrollment.
7. Pulmonary embolus within three weeks of enrollment as documented by computed tomography (CT) scan or nuclear scan.
8. Symptomatic cerebrovascular disease or a > 80% carotid stenosis.
9. Patients have moderate to severe aortic insufficiency without plans for correction during pump implantation surgery.
10. Patients with mechanical, animal or human tissue heart valves are excluded.
11. Severe right ventricular failure as defined by the anticipated need for right ventricular assist device (RVAD) support or extracorporeal membrane oxygenation (ECMO)at the time of HeartWare® LVAD screening/enrollment or right atrial pressure > 20 mmHg on multiple inotropes, right ventricular ejection fraction (RVEF) <15% or clinical signs including lower extremity edema, ascites or pleural effusions refractory to treatment with diuretics and two inotropic drugs.
12. Active, uncontrolled infection diagnosed by a combination of clinical symptoms and laboratory testing, including but not limited to, continued positive cultures, elevated temperature and white blood cell (WBC) count, hypotension, tachycardia, generalized malaise despite appropriate antibiotic, antiviral or antifungal treatment.
13. Uncorrected thrombocytopenia or generalized coagulopathy (e.g., platelet count < 100,000, INR > 1.6 or PTT > 2.5 times control in the absence of anticoagulation therapy).
14. Intolerance to anticoagulant or antiplatelet therapies or any other peri- or postoperative therapy that the investigator may administer based upon the patient's health status.
15. Serum creatinine greater than 3.0 times the upper limit of normal within 48 hours of study enrollment or requiring dialysis (does not include use of ultra-filtration for fluid removal).
16. All three listed liver enzymes [AST (SGOT), ALT (SGPT), or LDH] > 3 times upper limit of normal or a total bilirubin > 3 mg/dl within 24 hours of study enrollment, or biopsy proven liver cirrhosis or portal hypertension.
17. Pulmonary vascular resistance is unresponsive (fixed) to pharmacologic manipulation as demonstrated by a pulmonary artery systolic pressure exceeding 60mmHg in conjunction with any one of the three following variables:

    * Pulmonary vascular resistance is greater than 5 Woods Units or
    * Pulmonary vascular resistance index is greater than 6 Woods Units or
    * Transpulmonary gradient exceeds 16 to 20 mmHg
18. Patients requiring aortic, mitral, tricuspid or pulmonary valve replacements (including bioprosthetic valves) or left ventricular (LV) aneurysm resections.
19. Participation in any other study involving investigational drugs or devices.
20. Severe illness, other than heart disease, which would exclude cardiac transplantation.
21. Pregnancy.
22. Patient unwilling or unable to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2008-08; Primary Completion 2010-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Slaughter, MD, Principal Investigator — Jewish Hospital/Univ of Louisville; Keith Aaronson, MD, Principal Investigator — Univ of Michigan Medical Center
Locations (35):
- United States (35):
  - Mayo Clinic (Arizona), Phoenix, Arizona
  - Sharp Memorial Hospital, San Diego, California
  - Stanford University School of Medicine, Stanford, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida Gainesville, Gainesville, Florida
  - University of Miami / Jackson Memorial Hospital, Miami, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - IU Health Methodist, Indianapolis, Indiana
  - St. Vincent Health, Indianapolis, Indiana
  - Jewish Hospital - Rudd Heart and Lung Institute, Louisville, Kentucky
  - John Ochsner Heart & Vascular Institute, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic / St. Marys Hospital, Rochester, Minnesota
  - Washington University / Barnes Jewish Hospital, St Louis, Missouri
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundatiojn, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Texas Heart Institute, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Result] Aaronson KD, Slaughter MS, Miller LW, McGee EC, Cotts WG, Acker MA, Jessup ML, Gregoric ID, Loyalka P, Frazier OH, Jeevanandam V, Anderson AS, Kormos RL, Teuteberg JJ, Levy WC, Naftel DC, Bittman RM, Pagani FD, Hathaway DR, Boyce SW; HeartWare Ventricular Assist Device (HVAD) Bridge to Transplant ADVANCE Trial Investigators. Use of an intrapericardial, continuous-flow, centrifugal pump in patients awaiting heart transplantation. Circulation. 2012 Jun 26;125(25):3191-200. doi: 10.1161/CIRCULATIONAHA.111.058412. Epub 2012 May 22. PMID 22619284
- [Derived] Mahr C, McGee E Jr, Cheung A, Mokadam NA, Strueber M, Slaughter MS, Danter MR, Levy WC, Cheng RK, Beckman JA, May DM, Ismyrloglou E, Tsintzos SI, Silvestry SC. Cost-Effectiveness of Thoracotomy Approach for the Implantation of a Centrifugal Left Ventricular Assist Device. ASAIO J. 2020 Aug;66(8):855-861. doi: 10.1097/MAT.0000000000001209. PMID 32740343
- [Derived] Silvestry SC, Mahr C, Slaughter MS, Levy WC, Cheng RK, May DM, Ismyrloglou E, Tsintzos SI, Tuttle E, Cook K, Birk E, Gomes A, Graham S, Cotts WG. Cost-Effectiveness of a Small Intrapericardial Centrifugal Left Ventricular Assist Device. ASAIO J. 2020 Aug;66(8):862-870. doi: 10.1097/MAT.0000000000001211. PMID 32740129
- [Derived] Rahman F, McEvoy JW, Ohkuma T, Marre M, Hamet P, Harrap S, Mancia G, Rodgers A, Selvin E, Williams B, Muntner P, Chalmers J, Woodward M. Effects of Blood Pressure Lowering on Clinical Outcomes According to Baseline Blood Pressure and Cardiovascular Risk in Patients With Type 2 Diabetes Mellitus. Hypertension. 2019 Jun;73(6):1291-1299. doi: 10.1161/HYPERTENSIONAHA.118.12414. PMID 31030606
- [Derived] Teuteberg JJ, Slaughter MS, Rogers JG, McGee EC, Pagani FD, Gordon R, Rame E, Acker M, Kormos RL, Salerno C, Schleeter TP, Goldstein DJ, Shin J, Starling RC, Wozniak T, Malik AS, Silvestry S, Ewald GA, Jorde UP, Naka Y, Birks E, Najarian KB, Hathaway DR, Aaronson KD; ADVANCE Trial Investigators. The HVAD Left Ventricular Assist Device: Risk Factors for Neurological Events and Risk Mitigation Strategies. JACC Heart Fail. 2015 Oct;3(10):818-28. doi: 10.1016/j.jchf.2015.05.011. PMID 26450000
- [Derived] Birks EJ, McGee EC Jr, Aaronson KD, Boyce S, Cotts WG, Najjar SS, Pagani FD, Hathaway DR, Najarian K, Jacoski MV, Slaughter MS; ADVANCE Trial Investigators. An examination of survival by sex and race in the HeartWare Ventricular Assist Device for the Treatment of Advanced Heart Failure (ADVANCE) Bridge to Transplant (BTT) and continued access protocol trials. J Heart Lung Transplant. 2015 Jun;34(6):815-24. doi: 10.1016/j.healun.2014.12.011. Epub 2014 Dec 29. PMID 25813372
- [Derived] Goldstein DJ, Aaronson KD, Tatooles AJ, Silvestry SC, Jeevanandam V, Gordon R, Hathaway DR, Najarian KB, Slaughter MS; ADVANCE Investigators. Gastrointestinal bleeding in recipients of the HeartWare Ventricular Assist System. JACC Heart Fail. 2015 Apr;3(4):303-13. doi: 10.1016/j.jchf.2014.11.008. Epub 2015 Mar 11. PMID 25770405
- [Derived] Milano C, Pagani FD, Slaughter MS, Pham DT, Hathaway DR, Jacoski MV, Najarian KB, Aaronson KD; ADVANCE Investigators. Clinical outcomes after implantation of a centrifugal flow left ventricular assist device and concurrent cardiac valve procedures. Circulation. 2014 Sep 9;130(11 Suppl 1):S3-11. doi: 10.1161/CIRCULATIONAHA.113.007911. PMID 25200052
- [Derived] John R, Aaronson KD, Pae WE, Acker MA, Hathaway DR, Najarian KB, Slaughter MS; HeartWare Bridge to Transplant ADVANCE Trial Investigators. Drive-line infections and sepsis in patients receiving the HVAD system as a left ventricular assist device. J Heart Lung Transplant. 2014 Oct;33(10):1066-73. doi: 10.1016/j.healun.2014.05.010. Epub 2014 Jun 4. PMID 25087103
- [Derived] Najjar SS, Slaughter MS, Pagani FD, Starling RC, McGee EC, Eckman P, Tatooles AJ, Moazami N, Kormos RL, Hathaway DR, Najarian KB, Bhat G, Aaronson KD, Boyce SW; HVAD Bridge to Transplant ADVANCE Trial Investigators. An analysis of pump thrombus events in patients in the HeartWare ADVANCE bridge to transplant and continued access protocol trial. J Heart Lung Transplant. 2014 Jan;33(1):23-34. doi: 10.1016/j.healun.2013.12.001. Epub 2013 Dec 12. PMID 24418731
- [Derived] Slaughter MS, Pagani FD, McGee EC, Birks EJ, Cotts WG, Gregoric I, Howard Frazier O, Icenogle T, Najjar SS, Boyce SW, Acker MA, John R, Hathaway DR, Najarian KB, Aaronson KD; HeartWare Bridge to Transplant ADVANCE Trial Investigators. HeartWare ventricular assist system for bridge to transplant: combined results of the bridge to transplant and continued access protocol trial. J Heart Lung Transplant. 2013 Jul;32(7):675-83. doi: 10.1016/j.healun.2013.04.004. PMID 23796152

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 140 patients were enrolled at 30 sites into the study by giving written informed consent and were implanted with a HeartWare HVAD between August 18 2008 and February 23 2010.
Pre-assignment Details: This was a non randomized,open label,contemporaneously controlled trial. Pats. in the treatment arm were screened against the incl. & excl. criteria to determine eligibility to proceed to implant of the investigational device. Control Pats.contemporaneously entered into the INTERMACS (NCT00119834) database were selected using specified criteria.
Groups:
- HeartWare® VAS: Patients who received a HeartWare Ventricular Assist Device (HeartWare® VAS)
- Contemporaneous Control: Patients who received an FDA approved durable device for mechanically assisted support and enrolled into INTERMACS during the same enrollment period.
Period: Overall Study
Arm/Group | HeartWare® VAS | Contemporaneous Control
Started | 140 | 499
Completed | 140 | 499
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Contemporaneous Control: Patients who received an FDA approved durable device for mechanically assisted support and enrolled into INTERMACS (NCT00119834) during the same enrollment period.
- Total: Total of all reporting groups
Arm/Group | HeartWare® VAS | Contemporaneous Control | Total
Number analyzed (Participants) | 140 | 499 | 639
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (10.3) | 52.2 (12.2) | 52.2 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 120 | 159
  Male | 101 | 379 | 480
Region of Enrollment [Number; unit: participants]
  United States | 140 | 499 | 639
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 2.06 (0.28) | 2.07 (0.3) | 2.07 (0.29)
Blood Urea Nitrogen (BUN) [Mean (Standard Deviation); unit: mmol/L] | 9.12 (4.92) | 10.32 (7.48) | 10.06 (7.01)
Right Atrial Pressure (RAP) [Mean (Standard Deviation); unit: mmHg] | 11.14 (7.18) | 11.91 (6.79) | 11.84 (6.82)
Serum creatinine [Mean (Standard Deviation); unit: µmol/L] | 114.1 (39.1) | 121.9 (50) | 120.2 (47.9)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint is Success at 180 Days Which is Defined as Alive on the Originally Implanted HeartWare® LVAD or Transplanted or Explanted for Recovery. Patient Must Survive 60 Days Post-explant for Recovery to be Considered Successful.
Description: The primary endpoint is success at 180 days which is defined as alive on the originally implanted HeartWare® LVAD or transplanted or explanted for recovery. A patient must survive 60 days post-explant for recovery to be considered successful.
Time Frame: 180 days
Population: The primary effectiveness analyses was performed on the safety population, consisting of all enrolled subjects who received a Ventricular Assist Device (VAD).
Measure: Number; unit: Percentage of participants with success
Arm/Group | HeartWare® VAS | Contemporaneous Control
Number analyzed (Participants) | 140 | 497
Percentage of participants with success | 90.7 | 90.1

2. Secondary Outcome: Survival to 180 Days
Description: All subjects will be followed for date of death until 180 days.
Time Frame: 180 Days
Population: The secondary effectiveness analyses were performed on the safety population, consisting of all enrolled subjects who received a Ventricular Assist Device (VAD).
Measure: Number; unit: Percentage of participants with survival
Arm/Group | HeartWare® VAS | Contemporaneous Control
Number analyzed (Participants) | 140 | 499
Percentage of participants with survival | 94.3 | 91.2

3. Secondary Outcome: Incidence of Adverse Events, Neurocognitive Status and Unanticipated Adverse Device Effects
Description: Adverse events are only provided for patients who received a HeartWare Ventricular Assist Device (HeartWare® VAS). Adverse events as described by INTERMACS for the contemporaneous control population were not a part of the agreement for analysis and thus not provided by INTERMACS, and so not included in the Adverse Event Module and relevant Outcome Measures for comparison.
Time Frame: 180 Days
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | HeartWare® VAS
Number analyzed (Participants) | 140
percentage of patients
  Bleeding requiring reoperation | 17.1
  Infections - Local | 25.0
  Infections - Driveline | 12.1
  Infections - Sepsis | 11.4
  Neurologic Event-Ischemic Cerebrovascular accident | 7.1
  Neurologic Event-Hemorrhagic CVA | 4.3
  Neurologic Event - Transient Ischemic Attack(TIA)A | 4.3
  Right Heart Failure - requiring Inotropes | 16.0
  Right Heart Failure - requiring RVAD | 2.9
  Respiratory Dysfunction | 19.3
  Arterial Thromboembolism | 2.9
  Venous Thromboembolism | 6.4
  Renal Dysfunction | 5.7
  Hepatic Dysfunction | 2.9
  Hemolysis | 3.6

4. Secondary Outcome: Incidence of All Device Failures and Device Malfunctions
Description: The INTERMACS event device malfunction defined a failure of the HeartWare VAS as either pump failure or non-pump failure.
Time Frame: 180 Days
Population: as for outcome 2
Measure: Number; unit: Number of events
Arm/Group | HeartWare® VAS
Number analyzed (Participants) | 140
Number of events
  Pump Failure (exchange) | 7
  Non pump failure | 19

5. Secondary Outcome: Quality of Life Change From Baseline to 180 Days, as Measured by Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life for patients with congestive heart failure. It is a predictive tool that tracks how patients are doing if they have weakened heart muscle due to prior heart attacks, heart valve problems, viral infections, or other causes.
  The KCCQ's questions are used to calculate scores in ten domains:
  Physical Limitation, Symptom Stability, Frequency, Burden and Total Symptom. Social Limitation, Self-Efficacy, Quality of Life, and Clinical Summary. Overall Summary: a combined measure of all the above
  For each domain, the validity, reproducibility, responsiveness and interpretability have been independently established. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Baseline and 180 Days
Population: Number of participants with both baseline and 180 day data were used for this analysis of QOL.
Measure: Mean (Standard Deviation); unit: units on a KCCQ scale
Arm/Group | HeartWare® VAS
Number analyzed (Participants) | 70
units on a KCCQ scale | 30.94 (26.51)

6. Secondary Outcome: Change in Distance Walked in the 6-minute Walk Test Between Baseline and 180 Days
Description: The 6MWT is a simple test which does not require expensive equipment or advanced training for technicians. The test involves asking the patient to walk the longest distance possible in a set interval of 6 min, through a walking course (corridor) preferably 30-m long. The patient can stop or slow down at any time and then resume walking, depending on his/her degree of fatigue.
  A longer distance walked is indicative of a better outcome.
Time Frame: Baseline and 180 Days
Population: Number of participants with both baseline and 180 day data were used for this analysis of 6 minute walk distance.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | HeartWare® VAS
Number analyzed (Participants) | 74
meters | 150.14 (214.13)

7. Secondary Outcome: Quality of Life Change From Baseline to 180 Days, as Measured by EuroQoL EQ-5D
Description: The EQ-5D is a standardized instrument for use as a generic measure of the quality of health-related life and of health outcome.
  The EuroQoL EQ-5D is a descriptive system of health-related quality of life states consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of five responses. The responses record five levels of severity (no problems/slight problems/moderate problems/severe problems/extreme problems) within a particular EQ-5D dimension.
  Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Baseline and 180 Days
Population: Number of participants with both baseline and 180 day data were used for this analysis of QOL
Measure: Mean (Standard Deviation); unit: units on a EuroQol EQ-5D scale
Arm/Group | HeartWare® VAS
Number analyzed (Participants) | 72
units on a EuroQol EQ-5D scale | 29.53 (25.18)

ADVERSE EVENTS:
Time Frame: Adverse events were collected and are reported during the 180 day primary endpoint period.
Description: Treatment emergent adverse events are defined as events occurring after the skin incision for implantation of the pump. Adverse events that resulted in death, those assessed by the principal investigator as an SAE, any UADE, or those that met the definition of an INTERMACS event, were sent to the Clinical Events Committee with associated data.The Clinical Events Committee evaluated whether the event met the appropriate definition and determined the event's relationship to the device.
Arm/Group | HeartWare® VAS
Serious Adverse Events (participants affected / at risk) | 118/140
Other Adverse Events (participants affected / at risk) | 105/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HeartWare® VAS (N=140)
Cardiac disorders (Cardiac disorders) | 69 (99)
"Respiratory, thoracic and mediastinal disorders" (Respiratory, thoracic and mediastinal disorders) | 47 (78)
Infections and infestations (Infections and infestations) | 37 (56)
"Injury, poisoning and procedural complications" (Injury, poisoning and procedural complications) | 25 (34)
Nervous system disorders (Nervous system disorders) | 23 (32)
Gastrointestinal disorders (Gastrointestinal disorders) | 18 (29)
Vascular disorders (Vascular disorders) | 20 (26)
Investigations (Investigations) | 17 (21)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 12 (17)
Renal and urinary disorders (Renal and urinary disorders) | 14 (17)
General disorders and administration site conditions (General disorders) | 11 (12)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 9 (11)
Psychiatric disorders (Psychiatric disorders) | 5 (5)
Eye disorders (Eye disorders) | 3 (3)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 3 (3)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 3 (3)
Hepatobiliary disorders (Hepatobiliary disorders) | 2 (2)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 (1)
Immune system disorders (Immune system disorders) | 1 (1)
"Neoplasms benign, malignant and unspecified (including cysts and polyps)" (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Social circumstances (Social circumstances) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HeartWare® VAS (N=140)
"Respiratory, thoracic and mediastinal disorders" (Respiratory, thoracic and mediastinal disorders) | 46 (66)
Cardiac disorders (Cardiac disorders) | 37 (49)
Nervous system disorders (Nervous system disorders) | 32 (45)
Investigations (Investigations) | 22 (37)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 19 (23)
Gastrointestinal disorders (Gastrointestinal disorders) | 16 (20)
"Injury, poisoning and procedural complications" (Injury, poisoning and procedural complications) | 16 (17)
General disorders and administration site conditions (General disorders) | 12 (16)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 8 (11)
Vascular disorders (Vascular disorders) | 10 (11)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 9 (9)
Infections and infestations (Infections and infestations) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less